CLINICAL TRIAL: NCT06672666
Title: A Pilot Double-Blind Placebo-Controlled, Randomized, Safety, Efficacy, and Acceptability Trial of a Hemp-Derived Cannabidiol Extract for the Treatment of Anxiety
Brief Title: Use of CBD in the Treatment of Anxiety
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202301796
Record Dates: First submitted 2024-10-21; First posted 2024-11-04 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Anxiety; Generalized Anxiety Disorder; Sleep Problems
Keywords: Anxiety; CBD; Cannabidiol; Hemp-Derived Cannabidiol Extract; Generalized Anxiety Disorder; GAD; sleep
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder; Parasomnias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hemp Derived Cannabidiol Extract (Experimental): SunFlora's CBD Extract 50mg to 150mg titrated over 4 weeks
  Interventions: Drug: Hemp Derived Cannabidiol Extract
- Placebo (Placebo Comparator): Placebo substance to reflect same consistency as the experimental drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hemp Derived Cannabidiol Extract — Participants will be given the study drug in a titrated method of 50-150mgs per day for 4 weeks
  Other Names: SunFlora CBD Extract
  Arms: Hemp Derived Cannabidiol Extract
Drug: Placebo — Partcipants will be given placebo substance to be taken with titrated instructions that mimic IP dispensing method daily for 4 weeks
  Arms: Placebo

SUMMARY:
This study will examine the doses, safety, and test the preliminary efficacy of hemp-derived CBD product for improving anxiety symptoms and sleep disturbances among individuals with anxiety. A 4-week, randomized, double-blind, placebo-controlled trial will be conducted to determine the safety, tolerability, preliminary efficacy, and acceptability of 50 to 150 mg/day of CBD. The treatment period will consist of a two-week titration period followed by a 2- week maintenance period. In addition, the study seeks to examine whether changes in sleep disturbances precede changes in anxiety symptoms.

DETAILED DESCRIPTION:
Approximately one-third (33.1%) of Americans will experience an anxiety disorder at some point in their lifetime. Anxiety disorders are primarily treated with antidepressants or benzodiazepines, but unfortunately, many patients report a partial response or cannot tolerate the side effects of these medications, which include risk for abuse, cognitive impairment, and even death. The therapeutic potential of various compounds derived from the Cannabis sativa plant has generated considerable interest, particularly for managing neuropsychiatric disorders that have limited treatment options. Among these compounds, tetrahydrocannabinol (THC) and cannabidiol (CBD), have received significant attention. CBD has shown a unique pharmacological profile that lacks the potential for abuse associated with THC. Animal and small-scale human studies have demonstrated CBD's anxiolytic, antidepressant, panicolytic, and anticompulsive actions, however more research is needed to investigate the mechanisms of action and determine whether these products represent a safe and effective option for the treatment of anxiety. This study will examine the safety and test the preliminary efficacy of hemp-derived CBD product for improving anxiety symptoms and sleep disturbances among individuals with anxiety. A 4-week, randomized, double-blind, placebo-controlled trial will be conducted to determine the safety, tolerability, efficacy, and acceptability of 50 to 150 mg/day of CBD. The treatment period will consist of a two-week titration period followed by a 2- week maintenance period. Standardized questionnaires, blood, and urine exams will be used to comprehensively monitor adverse drug events. Clinical measurements will be performed to assess changes in anxiety and sleep quality. This study will also examine whether changes in sleep disturbances precede changes in anxiety symptoms. Participants will complete a comprehensive evaluation for the assessment of relevant medical history, and concomitant medication use. This study will provide information about the dosing and safety profile of a CBD hemp-based product and its major metabolites following single and multiple doses of a CBD extract among individuals with anxiety. In addition, the study will provide preliminary evidence of the independent and concomitant effects of CBD on anxiety symptoms and sleep patterns among individuals with anxiety and finally will assess the feasibility and acceptability of study procedures, including dosing, adherence to the study protocols, and the assessment of anxiety symptoms and sleep disturbances measurements over time.

ELIGIBILITY:
Inclusion Criteria:

* Any biological sex and ages 18 to 55 years old
* Willing and able to give informed consent for participation in the study
* Willing and able to comply with all study requirements, including willingness to donate blood during the study
* Meet diagnosis for moderate to severe anxiety based on a score of more than 14 in the Hamilton Anxiety Rating Scale (HAM-A)
* Subjects of childbearing potential should use two forms of highly effective contraception methods combined (e.g., barrier methods combined with Long-Acting Reversible Contraceptives) to be eligible for study participation.
* Normal clinical history and laboratory test

Exclusion Criteria:

* Pregnancy or breastfeeding
* Any history of suicidal behavior or any suicidal ideation in the past six months or at screening
* Any change in current SSRI, SNRI, or other non-benzo anxiolytic medication within six weeks of baseline visit.
* Active daily or almost daily (3+ days/week) use of cannabinoids or THC in the past month or any other illicit drug within the past 6 months
* Inability to refrain from using alcohol (4 or more drinks in one occasion or 3+ days/week), antiepileptics, antipsychotics, oral antifungals, verapamil, nitrofurantoin, or any other medication in drug classes, such as antibiotics, nonsteroidal anti-inflammatory drugs, herbal and dietary supplements, cardiovascular drugs, central nervous system agents, or antineoplastic drugs, inducing transaminase elevation based on the LiverTox database. 17,18
* Inability to adjust the doses of prescription medications displaying a narrow therapeutic index that are potentially impacted by concomitant cannabinoid use18,19.
* Inability to refrain from using acetaminophen, or topic antifungals on a regular basis (more than two times per week) over the course of the trial.
* Active use of benzodiazepines, opioids, and antihistamines or any other medication inducing lethargy and sedation, except for antidepressants, for which detailed information will be collected.
* History of liver disease or current liver disease or clinically significant elevation in serum liver chemistries at baseline (i.e., Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 times upper limit of normal (ULN) or alkaline phosphatase (ALP) >2 times ULN (or the baseline value if baseline is elevated); Total serum bilirubin >2.5 mg/dL with elevated AST, ALT or ALP; or International normalized ratio (INR) >1.5 with elevated AST, ALT or ALP).20
* Current substance use disorder
* Unstable medical or neurological condition
* Positive drug screen for substances of abuse
* Lifetime history of psychotic disorder, bipolar disorder, PTSD or OCD
* Psychotherapy newly instituted during the 6 weeks leading up to enrollment in the study. Subjects established in psychotherapy without change during the course of the study may participate.
* Severe depression symptoms in the past six months.
* Known or suspected hypersensitivity to cannabidiol or any other components in the extract.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Average CBD dose (mgs) used in the titration phase as reported in participant forms. | From enrollment to the end of titration phase at 2 weeks (Day 1 to Day 14).
  This trial will inform the dosing of a CBD hemp-based product and its major metabolites following single and multiple doses of a CBD extract (from 50 to 150 mg/day of CBD) among individuals with anxiety. The treatment period will consist of a two-week titration period followed by a 2- week maintenance period. Standardized questionnaires will be used to examine adherence to dosing protocol and potential changes due to side effects. During the titration phase, participants will be instructed to use an initial dosing of 50 mg/day in the morning progressively increasing 50 mg CBD/day before bedtime as tolerated by the individual participant, up to 150 mg/day by day 14. If a patient experiences mild side effects at doses at or higher than 50 mg daily, the investigators will monitor and may consider temporarily or permanently reducing the dose for the remainder of the study to the doses tolerated. Participants will report the daily doses used on a weekly basis in a dosing sheet.
Average CBD dose (mgs) used in the maintenance phase as indicated and reported in participant forms. | From week 2 to the end of maintenance phase at 4 weeks (Day 15 to Day 28)
  This trial will inform the dosing of a CBD hemp-based product and its major metabolites following single and multiple doses of a CBD extract (50 to 150 mg/day of CBD) among individuals with anxiety. The treatment period will consist of a two-week titration period followed by a 2- week maintenance period. Standardized questionnaires will be used to examine adherence to dosing protocol and potential changes due to side effects. During the maintenance phase, participants will stay at the optimal tolerated dose (between 50-150 mg) for two additional weeks. If a patient experiences mild side effects at doses at or higher than 50 mg daily, the investigators will monitor and may consider temporarily or permanently reducing the dose for the remainder of the study to the doses tolerated. Participants will report the daily doses used on a weekly basis in a dosing sheet.
Percentage of Severity of treatment-related adverse events based on the side effects/adverse events checklist, laboratory test, and self-report of unexpected ADE | From enrollment to the end of the study period at 12 weeks (Day 1 to Day 84)
  The safety and tolerability will be determined in eight-assessments conducted during a 12-week period, and based on the side effects/adverse events checklist, laboratory tests, and self-reports of unexpected adverse drug events (ADEs). The type of treatment-related adverse events based will be characterized based on those assessments. The side effects/adverse events will be categorized as: no ADEs, mild (i.e., no intervention required; no impact on activities of daily living), moderate (minimal, local, or non-invasive intervention indicated; moderate impact on activities of daily living) or severe (i.e., significant symptoms requiring invasive intervention; subject seeks medical attention, needs major assistance).
Percentage of patients reporting Drug-Induced Liver Injury based on liver chemistries | From enrollment to the end of the study period at 12 weeks (Day 1 to Day 84).
  In this study, patients are going to be followed for 84 days after treatment initiation, with serum liver chemistries assessments at baseline, and in four subsequent visits (visits 3, 5, 6 and 8), with the last serum liver chemistries 49 days after the last doses. The result is reported as the number of participants that had a clinically significant clinically significant elevation in serum liver chemistries (i.e., Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 times upper limit of normal (ULN) or alkaline phosphatase (ALP) >2 times ULN, Total serum bilirubin >2.5 mg/dL with elevated AST, ALT or ALP; or International normalized ratio (INR) >1.5 with elevated AST, ALT or ALP.
Percentage of severity of depression symptoms based on the Patient Health Questionnaire-9 | From enrollment to the end of the study period at 12 weeks (Day 1 to Day 84).
  The Patient Health Questionnaire-9 is a 9-item scale useful for the assessment of the presence and severity of depressive symptom, and a possible depressive disorder. Each of the nine items reflects a DSM-5 symptom of depression. PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively.
Percentage of participants reporting suicidal ideation and behavior based on the Columbia Suicide Severity Rating Scale | From enrollment to the end of the study period at 12 weeks (Day 1 to Day 84).
  The Columbia Suicide Severity Rating Scale (C-SSRS) is a 6-item scale that assesses suicidal ideation and behavior by helping to identify specific behaviors that may be indicative of an individual's intent to kill oneself. Four constructs are measured, including: severity of ideation, intensity of ideation, behavior and lethality.

SECONDARY OUTCOMES:
Change in anxiety symptoms scores based on the Hamilton Anxiety Rating Scale. | From enrollment to the end of treatment at 4 weeks
  This study will provide preliminary evidence of the independent and concomitant effects of CBD on anxiety symptoms among individuals with moderate to severe anxiety. Anxiety symptoms will be assessed over the 12-week period using the Hamilton Anxiety Rating Scale (HAM-A). This scale consists of 14 symptom-defined elements, and caters for both psychological (e.g., fears, anhedonia) and somatic (e.g., tachycardia, chest tightness) symptoms. Each item is scored on a basic numeric scoring of 0 (not present) to 4 (severe). HAM-A score ranges are: mild anxiety = 8-14; moderate = 15-23; severe 24 or more. Scores below 8 were considered to represent no/minimal anxiety. For this study the HAM-A test will be conducted during eight assessments in the 12-week study period.
Change in perceived severity of anxiety symptoms and functionality based on the Clinical Global Impression. | From enrollment to the end of treatment at 4 weeks
  This study will assess the change in perceived severity of anxiety symptoms and functionality based on the Clinical Global Impression (CGI). The CGI is a 3-item scale that assesses the patient's functioning prior to and after initiating medication in trials which is an important part of the study process. Its 3 items assess, 1) Severity of Illness (CGI-S), 2) Global Improvement (CGI-I), and 3) Efficacy Index (CGI-E, which is a measure of treatment effect and side effects specific to drugs that were administered). For this study the CGI test will be conducted during eight assessments in the 12-week study period.
Change in generalized anxiety symptoms and severity based on the Generalized Anxiety Disorder 7 scale | From enrollment to the end of treatment at 4 weeks.
  This study will provide preliminary evidence of the independent and concomitant effects of CBD on generalized anxiety symptoms among individuals with moderate to severe anxiety using the Generalized Anxiety Disorder 7 (GAD 7). This 7-items scale with strong criterion validity is useful for identifying probable cases of GAD and assessing its severity. Increasing scores on the GAD-7 are strongly associated with multiple domains o symptoms will be assessed over the 12-week study period.
Change in sleep quality and disturbances based on the Pittsburgh Sleep Quality Index (PSQI): | From enrollment to the end of treatment at 4 weeks.
  This study will provide preliminary evidence of the independent and concomitant effects of CBD on improving sleep based on the Pittsburgh Sleep Quality Index (PSQI). This 19-item scale assesses sleep quality and disturbances over a 1-week time interval. The items generate seven "component" scores, including: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
Changes in insomnia symptoms based on the Insomnia Severity Index. | From enrollment to the end of treatment at 4 weeks.
  This study will provide preliminary evidence of the independent and concomitant effects of CBD on improving sleep based on the following self-report assessments. Changes in insomnia symptoms will be estimated using the Insomnia Severity Index (ISI). This 7-item scale assesses the severity of sleep-onset and sleep maintenance difficulties (both nocturnal and early morning awakenings), satisfaction with current sleep pattern, interference with daily functioning, noticeability of impairment attributed to the sleep problem, and degree of distress or concern caused by the sleep problem. Each item is rated on a 0-4 scale and the total score ranges from 0 to 28. A higher score suggests more severe insomnia.
Average of acceptability to study procedures score based on feasibility and acceptability study forms | From enrollment to the end of the study period at 12 weeks (Day 1 to Day 84).
  This study will collect data on the acceptability of the study procedures which examine adherence to the study protocols, including acceptability of study procedures (e.g., adjustment of daily activities to participate in the study and levels of engagement) using standardized forms designed by the research team and based on prior studies. The form is a 7-point 15 item scale that will be conducted during six in-person and two phone assessments.
Percentage of participants reporting levels of adherence to study procedures based on feasibility and acceptability study forms | From enrollment to the end of the study period at 12 weeks (Day 1 to Day 84).
  This study will collect weekly data on the feasibility and acceptability (F&A) form of the study procedures which examine levels (low, middle and high) of adherence to the study protocols, including missing doses and adherence to procedures (e.g., completion of lab and questionnaire assessments, adherence to recommended doses) using a 15-item standardized form designed by the research team and based on prior studies. Patients will be asked to return unused medications every other week when the new product is dispensed. The research team will check the returned medications against the usage recorded. Any discrepancies will be discussed with the patient and documented accordingly within the patient's source documents.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
The approved Informed Consent Form restricts the sharing of individual data.